CLINICAL TRIAL: NCT03667300
Title: Evogliptin Versus Linagliptin for the Effect on Albuminuria in Patients With Type 2 Diabetes and Renal Insufficiency: a Multicenter, Randomised, Double-blind, Active-controlled, Non-inferiority Trial
Brief Title: Effect of Evogliptin on Albuminuria in Patients With Type 2 Diabetes and Renal Insufficiency
Acronym: DA1229
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jae Hyeon Kim, MD, PhD, Professor / Division of Endocrinology and metabolism, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016-08-144
Record Dates: First submitted 2018-02-20; First posted 2018-09-12 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Type2 Diabetes Mellitus; Albuminuria; Renal Insufficiency
Keywords: Type2 Diabetes Mellitus; Intervention; Albuminuria
MeSH Terms: conditions — Albuminuria; Renal Insufficiency | interventions — 4-(3-amino-4-(2,4,5-trifluorophenyl)butanoyl)-3-(tert-butoxymethyl)piperazin-2-one; Linagliptin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Evogliptin Group (Active Comparator): Intervention group will take daily evogliptin 5mg per oral, not linagliptin 5mg per oral
  Interventions: Drug: Evogliptin
- Linagliptin Group (Active Comparator): Control group will take daily linagliptin 5mg per oral, not evogliptin 5mg per oral
  Interventions: Drug: Linagliptin

INTERVENTIONS:
Drug: Evogliptin — This group will take daily evogliptin 5mg per oral, not linagliptin.
  Other Names: Suganon
  Arms: Evogliptin Group
Drug: Linagliptin — This group will take daily linagliptin 5mg per oral, not evogliptin
  Other Names: Trajenta
  Arms: Linagliptin Group

SUMMARY:
In this multi-center, randomized, double-blind, active-controlled, phase II non-inferiority study, we aimed to test the non-inferiority of evogliptin vs linagliptin in terms of reduction of albuminuria at week 24 from baseline in patients with type 2 diabetes having renal insufficiency.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, active-controlled, phase II non-inferiority study. Evogliptin (Trade name, Suganon) is a new, novel dipeptidyl peptidase-4 (DPP4) inhibitor which reveals a favorable results on glucose-lowering effect in patients with diabetes. However, its effect on renal function in patients with diabetes has been uncertained. To compare the effect of evogliptin and linagliptin on the reduction of albuminuria, we will recruit a total of 210 patients with Type 2 diabetes and renal insufficiency and allocate the participants into evogliptin group and linagliptin group with a ratio of 1:1 after radomization from 10 hospitals. After the oral administration of evogliptin 5mg per day or linagliptin 5mg per day for 24 weeks, the percent change of urine albumin-to-creatinine ratio (UACR) at Week 24 and at baseline will be measured as a primary endpoint. In addition, the percent changes of UACR, hemoglobin A1c, Cystatin-C, Nephrin, N-acetyl-beta-D-glucosaminidase (NAG), glycated albumin, estimated glomerular filtration rate (eGFR) between baseline and Week 12 or Week 24 will be studied as secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 20 years or older diagnosed with type 2 diabetes.
* subjects having a level of glycated hemoglobin (HbA1c) 7.0% or more, and 10% or less.
* subjects having urine albumin to creatinine ratio (UACR) 30 ug/mg or more, and 3000 ug/mg or less.
* subjects having estimated glomerular filtration rate (eGFR) 30 or more.
* subjects who had taken angiotensin II receptor blocker(ARB) or angiotensin-converting enzyme(ACE) inhibitors for more than 4 weeks.
* subjects having body mass index (BMI) 20kg/m2 or more, 40 kg/m2 or less.
* subjects who entirely understood all the process of clinical study protocol and voluntarily take part in the study and agree to follow rule of the study.

Exclusion Criteria:

* subjects having type 1 diabetes, secondary diabetes, or gestational diabetes
* subjects who had a history of surgery of resection of more than a half length of stomach or intestine.
* subjects having more than three-fold higher levels of Aspartate Transaminase(AST) or Alanine Transaminase(ALT) than upper normal limit.
* subjects who had taken Dipeptidyl Peptidase4(DPP4)-inhibitor or glucagon-like peptide-1(GLP-1) analogue within 8 weeks prior to screening.
* subjects who had taken oral triple hypoglycemic agents within 8 weeks prior to screening
* subjects taking strong cytochrome P450 3A4(CYP3A4) inhibitors or strong cytochrome P450 3A4(CYP3A4) inducers
* subjects who are pregnants or breast feeding givers.
* subjects who are unsuitable for clinical trial participation based on clinical laboratory test results or other reasons (e.g. taking chemotherapy or radiation for treatment for cancers).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2017-03-16 (Actual); Primary Completion 2019-05-14 (Actual); Study Completion 2019-05-14 (Actual)

PRIMARY OUTCOMES:
UACR percent change at Week 24 | Week 24
  Percentage change in urine albumin-to-creatinine ratio (UACR) after 24 weeks compared to baseline (%)

SECONDARY OUTCOMES:
UACR change at Week 24 (%) | Week 24
  Change in urine albumin-to-creatinine ratio (UACR) after 24 weeks compared to baseline (%)
UACR change at Week 12 | Week 12
  Change in urine albumin-to-creatinine ratio (UACR) after 12 weeks compared to baseline (mg/g
HbA1c change at Week 24 | Week 24
  Change in glycated hemoglobin after 24 weeks compared to baseline
HbA1c change at Week 12 | Week 12
  Change in glycated hemoglobin after 12 weeks compared to baseline
HbA1c less than 6.5% at Week 24 | Week 24
  proportion of parcipitants having glycated hemoglobin less than 6.5% after 24 weeks
HbA1c less than 6.5% at Week 12 | Week 12
  proportion of participants having glycated hemoglobin less than 6.5% after 12 weeks
HbA1c less than 7.0% at Week 24 | Week 24
  proportion of participants having glycated hemoglobin less than 7.0% after 24weeks
HbA1c less than 7.0% at Week 12 | Week 12
  proportion of participants having glycated hemoglobin less than 7.0% after 12 weeks
NAG (N-acetyl-β-D-glucosaminidase) change at Week 24 | Week 24
  Change in NAG (N-acetyl-β-D-glucosaminidase) after 24 weeks compared to baseline (U/L)
NAG (N-acetyl-β-D-glucosaminidase) change at Week 12 | Week 12
  Change in NAG (N-acetyl-β-D-glucosaminidase) after 12 weeks compared to baseline (U/L)
Cystatin-C change at Week 24 | Week 24
  Change in urinary Cystatin-C after 24 weeks compared to baseline (mg/L)
Cystatin-C change at Week 12 | Week 12
  Change in urinary Cystatin-C after 12 weeks compared to baseline (mg/L)
Nephrin change at Week 24 | Week 24
  Change in Nephrin after 24 weeks compared to baseline (ug/g cr)
Nephrin change at Week 12 | Week 12
  Change in Nephrin after 12 weeks compared to baseline (ug/g cr)
Glycated albumin change at Week 24 | Week 24
  Change in Glycated albumin after 24 weeks compared to baseline (%)
Glycated albumin change at Week 12 | Week 12
  Change in Glycated albumin after 12 weeks compared to baseline (%)
eGFR at Week 24 | Week 24
  Change in estimated glomerular filtration rate based on Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) method after 24 weeks compared to baseline (mL/min)
eGFR change at Week 12 | Week 12
  Change in estimated glomerular filtration rate based on Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) method after 12 weeks compared to baseline (mL/min)

CONTACTS AND LOCATIONS:
Overall Officials: Jae Hyeon Kim, MD PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No